

Title: A Phase 1, Open-label Study of Niraparib as Single Agent in Patients With Advanced Solid Tumors

NCT Number: NCT03497429

Statistical analysis plan Approve Date: 03-APR-2019

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).



### STATISTICAL ANALYSIS PLAN

# Applicable Terms of Use tie PLAN Araparib-1001 Araparib as Single Agent is need Solid Tumors PHASE 1 Version: 2nd Date: 03 April 2019 I on: Protocol Version: Initial version officel Date: 18 January 2018 A Phase 1, Open-label Study of Niraparib as Single Agent in Patients

Prepared by:

Protocol Version: Initial version
Protocol Date: 18 January 2018

Property of Takeda. For non-commercial use only and subject to the applicable Tames of use

# 2.0 TABLE OF CONTENTS

| | 1.1 | A | approval Signatures | 2 |
|---|---|---|---|---|
| 2.0 | | TAB | LE OF CONTENTS | 3 |
| 3.0 | | LIST | OF ABBREVIATIONS | 5 |
| 4.0 | | OBJI | ECTIVES | 6 |
| | 4.1 | p | rimary Objectives | 6 |
| | 4.2 | S | econdary Objectives | 6 |
| | 4.3 | A | Additional Objectives | 6 |
| | 4.4 | S | econdary Objectives | 6 |
| 5.0 | | ANA | LYSIS ENDPOINTS | 7 |
| | | 5.1.1 | LYSIS ENDPOINTS Primary Endpoints Secondary Endpoints Additional Endpoints ERMINATION OF SAMPLE SIZE | 7 |
| | | 5.1.2 | Secondary Endpoints | 7 |
| | | 5.1.3 | Additional Endpoints | 7 |
| 6.0 | | DET | ERMINATION OF SAMPLE SIZE | 8 |
| 7.0 | | | | |
| | 7.1 | C | Seneral Principles Study Definitions Definition of Study Visit Windows | 9 |
| | | 7.1.1 | Study Definitions | 9 |
| | | 7.1.2 | Definition of Study Visit Windows | 9 |
| | | 7.1.3 | Conventions for Missing Adverse Event Dates | 10 |
| | | 7.1.4 | Conventions for Missing Concomitant Medication Dates | 10 |
| | 7.2 | A | nalysis Sets<br>Disposition of Subjects | 10 |
| | 7.3 | Г | | |
| | | 7.3.1 | Study Information | 11 |
| | | 7.3.2 | Screen Failures | 11 |
| | | 7.3.3 | Subject Eligibility | 11 |
| | | 7.3.4 | Disposition of Subjects | 12 |
| | | 7.3.5 | Protocol Deviations and Analysis Sets | 12 |
| | 7.4 | Ę | Demographic and Other Baseline Characteristics | 13 |
| | 7.5 | (S) | Medical History and Concurrent Medical Conditions | 14 |
| | 7.6 | N | Medication History and Concomitant Medications | 15 |
| X | 7.7 | S | tudy Drug Exposure and Compliance | 15 |
| O. | 7.8 | E | fficacy Analysis | 16 |
| 1 | | 7.8.1 | Primary Efficacy Endpoint(s) | 16 |
| | | 7.8.2 | Secondary Efficacy Endpoint(s) | 16 |
| | | 7.8.3 | Additional Efficacy Endpoint(s) | 16 |

| 7.8.4 | Statistical/Analytical Issues | | 16 |
|---|---|---|---|
| | Pharmacokinetic/Pharmacodynamic Analysis | | |
| 7.9.1 | - | | |
| 7.9.2 | | | |
| 7.10 C | Other Outcomes | | 47.7 |
| 7 11 C | lafaty Analyzaia | | 10 |
| 7.11. | 1 Adverse Events | 20/4 | 19 |
| 7.11. | 2 Clinical Laboratory Evaluations | ::00 | 22 |
| 7.11. | 3 Vital Signs and Weight | | 23 |
| 7.11. | 4 12-Lead ECGs | | 23 |
| 7.11. | 1 Adverse Events | illo | 23 |
| 7.12 In | nterim Analysis | NO. | 23 |
| 7.13 C | Changes in the Statistical Analysis Plan | | 23 |
| 8.0 REF | ERENCES | 16, | 25 |
| | | 350 | |
| LIST OF IN | nterim Analysis Changes in the Statistical Analysis Plan ERENCES | | |
| EIST OF IN | VELOCIE II I I I I | | 10 |
| Table 7.a | Visit Window of Clinical Laboratory Tes | st | 10 |
| | , c. C | | |
| LIST OF IN | N-TEXT FIGURES | | |
| Figure 4.a | Schematic of Study Design | | 6 |
| S | | | |
| | Schematic of Study Design | | |
| | CO. | | |
| | ₹0, | | |
| 20 | | | |
| 160. | | | |
| 1 SIL | | | |
| Ex | | | |
| OCI | | | |
| OKOK | | | |
| Property of Lakeds | | | |

### 3.0 LIST OF ABBREVIATIONS

ΑE adverse event

ALT alanine aminotransferase AML acute myeloblastic leukemia

aPTT activated partial thromboplastin time

AST aspartate aminotransferase

AUC24 area under the plasma concentration-time curve

**BRCA** breast cancer (gene)

C24 plasma concentration at 24 hrs after last dose

maximum observed concentration Cmax

Cmin minimum observed concentration at multiple dose

CR complete response

**CRO** contract research organization CTcomputed tomography CYP cytochrome P450 DLT dose-limiting toxicity DNA deoxyribonucleic acid

Eastern Cooperative Oncology Group **ECOG** eCRF electronic case report form

(United States) Food and Drug Administration **FDA** 

**FSH** follicle stimulating hormone **GCP** Good Clinical Practice hepatitis B core antibody **HBcAb** hepatitis B surface antibody **HBsAb** hepatitis B surface antigen **HBsAg** 

hepatitis B virus **HBV HCV** hepatitis C virus

la: Fot vou. hepatitis C virus antibody **HCVAb** HIV human immunodeficiency virus HRD homologous recombination deficiency

**ICF** informed consent form

**ICH** International Council for Harmonisation of Technical Requirements for

Pharmaceuticals for Human Use

MedDRA Medical Dictionary for Regulatory Activities

ORR ? overall response rate

R(AUC24) accumulation ratio based on AUC24 R(Cmax) accumulation ratio based on Cmax Tmax time of first occurrence of C<sub>max</sub> TEAE treatment-emergent adverse event

### 4.0 OBJECTIVES

### 4.1 Primary Objectives

To evaluate the safety and tolerability of niraparib administered orally QD to Japanese patients with advanced solid tumors.

### 4.2 Secondary Objectives

To evaluate the pharmacokinetics of niraparib administered orally QD to Japanese patients with advanced solid tumors.

### 4.3 Additional Objectives

To evaluate the anti-tumor activity of niraparib administered orally QD to Japanese patients with advanced solid tumors

### 4.4 Study Design

This study is a phase 1, open-label, non-randomized, cohort-based, dose-escalation study to establish the safety and tolerability of niraparib in Japanese patients with advanced solid tumors. A total of 6 to 12 patients are treated with 200 mg QD (Cohort 1) or 300 mg QD (Cohort 2).

Niraparib will be administered QD, continuously for 21 days in Cycle 1. There will be no drug holiday. Niraparib will be administered QD, continuously in 21-day cycles from Cycle 2 onward. Episodes of DLT within the first 21 days of Cycle 1 are used to decide whether to escalate the dose. Subjects will receive niraparib under impatient hospitalization (hospitalization from Cycle 1 Day 1 to Cycle 1 Day 8 will be mandatory) and monitored for DLTs. Escalation to the next dose level does not occur until the results of safety measurements from Cycle 1 have been obtained and reviewed. The overview of study design is shown in Figure 4.a.





### 5.0 ANALYSIS ENDPOINTS

### 5.1.1 Primary Endpoints

- The number and percentage of subjects with DLTs during Cycle 1.
- The number and percentage of subjects with TEAEs.
- The number and percentage of subjects with Grade 3 or higher TEAEs.
- The number and percentage of subjects with serious TEAEs.
- The number and percentage of subjects who discontinued the study drug because of TEAEs.

# 5.1.2 Secondary Endpoints

• PK parameters of niraparib on Cycle 1 Day 1 and Day 21: Cmax, Tmax and AUC24.

### 5.1.3 Additional Endpoints

- Overall response rate (ORR) (complete response [CR] + partial response [PR]) as measured by the RECIST guidelines.
- Laboratory safety assessments, Eastern Cooperative Oncology Group (ECOG) performance status, electrocardiograms (ECGs) and vital signs.
- PK parameters of a metabolite, M1, on Cycle 1 Day 1 and Day 21: Cmax, Tmax and AUC24.

  PK parameters of a metabolite, M1, on Cycle 1 Day 1 and Day 21: Cmax, Tmax and AUC24.

  PK parameters of a metabolite, M1, on Cycle 1 Day 1 and Day 21: Cmax, Tmax and AUC24.

  PK parameters of a metabolite, M1, on Cycle 1 Day 1 and Day 21: Cmax, Tmax and AUC24.

Properly of Takeda, For non-confinercial use only and subject to the applicable of the property of takeda, For non-confinercial use only and subject to the applicable of the property of takeda.

### 7.0 METHODS OF ANALYSIS AND PRESENTATION

### 7.1 General Principles

### 7.1.1 Study Definitions

The following definitions and calculation formulas will be used.

- Treatment-emergent adverse event (TEAE): Adverse events that occur after administration of the first dose of study drug and through 28 days after the last dose of study drug.
- Pretreatment event (PTE): Any untoward medical occurrence in a clinical investigation subject who has signed informed consent to participate in a study but prior to administration of study drug.
- Descriptive statistics: Number of subjects, mean, standard deviation, maximum, minimum, and quartiles
- Dose: Initial dose level of 200 mg for Niraparib, Initial dose level of 300 mg for Niraparib.
- Group: Initial dose level of 200 mg for Niraparib, Initial dose level of 300 mg for Niraparib.
- Coefficient of variation (CV) (%): Standard deviation / mean \* 100.

### 7.1.2 Definition of Study Visit Windows

When calculating Study Day relative to a reference date (ie, date of first dose [Day 1]), if the date of the observation is on the same date or after the reference date, it will be calculated as: date of observation - reference date + 1; otherwise, it will be calculated as: date of observation - reference date. Hence, reference day is always Day 1 and there is no Day 0.

All evaluable data (ie, non-missing data) will be handled according to the following rules.

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Study Day to the scheduled Study Day will be used. If there are two observations equidistant to the scheduled Study Day, the later observation will be used.

Table 7.a Visit Window of Clinical Laboratory Test

| Visit | Scheduled S<br>(day | | Time Interval (days)<br>Study Day |
|---|---|---|---|
| Cycle 1, Day 1(Predose) | Study Day: | 1 | -7 to 1 |
| Cycle 1, Day 8 | Study Day: | 8 | 5 to 11 |
| Cycle 1, Day 15 | Study Day: | 15 | 12 to 18 |
| Cycle 2, Day 1 | Study Day: | 22 | 19 to 25 |
| Cycle 2, Day 8 | Study Day: | 29 | 26 to 32 |
| Cycle 2, Day 15 | Study Day: | 36 | 33 to 39 |
| Cycle (n) (Cycle 3 and thereafter), Day 1 | Study Day: | 21(n - 1) + 1 | 21(n - 1) - 2 to 21(n - 1) + 4 |
| Cycle (n) (Cycle 3 and<br>thereafter), Day 8 | Study Day: | 21(n - 1) + 8 | 21(n - 1) + 5 to 21(n - 1) + 11 |

# 7.1.3 Conventions for Missing Adverse Event Dates

Not applicable.

# 7.1.4 Conventions for Missing Concomitant Medication Dates

Not applicable.

### 7.2 Analysis Sets

• Safety analysis set:

Patients who receive at least 1 dose of study drug.

• Pharmacokinetic analysis set:

Patients with sufficient dosing and PK measurement data to reliably estimate 1 or more PK parameters.

• DLT-evaluable set:

Patients who have received at least 80% of planned doses of niraparib in Cycle 1 (for at least 17 days out of 21 days) unless interrupted by study drug-related toxicities and have sufficient follow-up data considered by sponsor and investigator to determine whether DLT occurred.

Response-evaluable set:

Patients who receive at least 1 dose of study drug, have sites of measurable disease at baseline, and have at least 1 postbaseline disease assessment.

### 7.3 **Disposition of Subjects**

### **Study Information** 7.3.1

Analysis Set:

All Subjects Who Signed the Informed Consent Form

Analysis Variable(s):

Date First Subject Signed Informed Consent Form

Date of Data Cutoff

MedDRA Version

WHO Drug Version

SAS Version Used for Creating the Datasets

Analytical Method(s):

(1) Study Information

### 7.3.2 Screen Failures

Analysis Set:

All Subjects Who Did Not Enter the Treatment Period

Analysis Variable(s):

Age (years)

Gender

Analytical Method(s):

(1) Screen Failures

. Osed for Creating the Datasets
.ethod(s):
Study Information
Study information shown in the analysis variables section will be provided.
en Failures

bjects Who Did Not Enter the Treatment Period
ble(s):
urs)
[Male, Female]
d(s):
Failures
bey die\* Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided.

# 7.3.3 Subject Eligibility

Analysis Set:

All Subjects Who Signed the Informed Consent Form

All Subjects V
Analysis Variable(s):
Eligibilit

**Eligibility Status** 

[Eligible for Entrance into the Treatment Period, Not Eligible for Entrance into the Treatment Period]

Primary Reason for Subject Not Being Eligible

[Death, Adverse Event, Protocol Deviation, Study Terminated by Sponsor, Withdrawal by Subject, Lost to Follow-up, Screen Failure, Other]

### Analytical Method(s):

(1) Eligibility for Entrance into the Treatment Period

Frequency distributions will be provided. When calculating percentages for the primary reasons for subject not being eligible, the total number of ineligible subjects nd subject to the appl will be used as the denominator.

### 7.3.4 Disposition of Subjects

Analysis Set:

All Subjects Who Entered the Treatment Period

Analysis Variable(s):

Study Drug Administration Status

[Ongoing, Discontinued]

Reason for Discontinuation of Study Drug Administration

[Death, Adverse Event, Protocol Deviation, Progressive Disease, Study Terminated by Sponsor, Pregnancy, Withdrawal by Subject, Lost to Follow-up, Otherl

### Analytical Method(s):

(1) Disposition of Subjects

Frequency distributions will be provided by dose and overall. When calculating percentages for the reasons for discontinuation, the total number of subjects who discontinued treatment will be used as the denominator.

# **Protocol Deviations and Analysis Sets**

### 7.3.5.1 Protocol Deviations

Analysis Set:

All Subjects Who Entered the Treatment Period

Analysis Variable(s):

Significant Protocol Deviation

[Entry Criteria, Concomitant Medication, Procedure Not Performed Per Protocol, Study Medication, Withdrawal Criteria, Major GCP Violations]

### Analytical Method(s):

(1) Protocol Deviations

category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the same category will be counted only once.

alysis Sets

t: to the applicable

### 7.3.5.2 Analysis Sets

Analysis Set:

All Subjects Who Entered the Treatment Period

Analysis Variable(s):

Handling of Subjects

[Categories are based on the specifications in Subject Evaluability List]

Analysis Sets

Safety Analysis Set [Included] Pharmacokinetic Analysis Set [Included] [Included] DLT-evaluable Set Response-evaluable Set [Included]

Analytical Method(s):

- (1) Subjects Excluded from Analysis Sets
- (2) Analysis Sets

Frequency distributions will be provided by dose for (1), and by dose and overall for (2). For (1), a subject who has several reasons for exclusion will be counted once in each appropriate category. A subject who has several reasons for exclusion that can be classified into the same category will be counted only once.

### 7.4 **Demographic and Other Baseline Characteristics**

Analysis Set:

Safety Analysis Set

Analysis Variable(s):

Age (years)

[Male, Female] Gender

Height (cm)

Weight (kg)

BMI  $(kg/m^2)$ 

[American Indian or Alaska Native, Asian, Black or African American, Race Native Hawaiian or Other Pacific Islander, White]

ECOG performance status [0, 1, 2, 3, 4]

[Adrenal cancer, Breast cancer, Cervical cancer, Colorectal cancer Diagnosis Endometrial cancer, Gastric cancer, Head and neck cancer, Liver cancer, Malignant Subject to the ap melanoma, Non small cell lung cancer, Ovarian cancer, Pancreatic cancer, Prostatic cancer, Small cell lung cancer, Other]

Prior Surgery/Procedure [Yes, No]

Prior Radiation Therapy [Yes, No]

**BRCA1** Mutant [Yes, No, Unknown]

**BRCA2 Mutant** [Yes, No, Unknown]

Analytical Method(s):

(1) Summary of Demographics and Baseline Characteristics

Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided by dose and overall.

### **Medical History and Concurrent Medical Conditions** 7.5

Analysis Set:

Safety Analysis Set

Analysis Variables:

Medical History

Concurrent Medical Conditions

Analytical Methods:

- (1) Medical History by System Organ Class and Preferred Term
- (2) Concurrent Medical Conditions by System Organ Class and Preferred Term

Frequency distributions will be provided by dose and overall. MedDRA dictionary will be used for coding. Summaries will be provided using SOC and PT, where SOC will be sorted alphabetically and PT will be sorted in decreasing frequency. A subject with multiple occurrences of medical history or concurrent medical condition within a SOC will be counted only once in that SOC. A subject with multiple occurrences of medical history or concurrent medical condition within a PT will be counted only once in that PT.

### 7.6 **Medication History and Concomitant Medications**

Analysis Set:

Safety Analysis Set

Analysis Variables:

Prior Anticancer Drug Therapy

**Concomitant Medications** 

Analytical Methods:

- (1) Prior Anticancer Therapy by Preferred Medication Name.
- in Phicable Terms of Use (2) Concomitant Medications That Started and Stopped Prior to Baseline by Preferred Medication Name.
- (3) Concomitant Medications That Started Prior to and Were Ongoing at Baseline as well as Those That Started After Baseline by Preferred Medication Name.

Frequency distributions will be provided by dose and overall. WHO Drug dictionary will be used for coding. Summaries will be provided using preferred medication names and sorted in decreasing frequency based on the number of reports. A subject who has been administered several medications with the same preferred medication name will be counted only once for that preferred medication name.

### Study Drug Exposure and Compliance 7.7

Analysis Set:

DLT-evaluable Set

Safety Analysis Set

Analysis Variable(s):

Treatment Compliance at Cycle1 (%)

 $[Min \le - < 80, 80 \le - < = Max]$ 

Days on Treatment

Number of Cycles

Analytical Method(s):

(1) Study Drug Exposure and Compliance

Frequency distributions and descriptive statistics for continuous variables will be provided by dose and overall.

### 7.8 **Efficacy Analysis**

### 7.8.1 **Primary Efficacy Endpoint(s)**

Not applicable.

### 7.8.2 Secondary Efficacy Endpoint(s)

Not applicable.

### 7.8.3 Additional Efficacy Endpoint(s)

Analysis Set:

Response-Evaluable Analysis Set

Analysis Variables:

**ORR** 

[CR, PR, SD, PD, NE] Overall Response

Analytical Methods:

(1) Primary Analysis

and subject to the applicable Terms of Use applicable Terms of Use For ORR, point estimate and the 2-sided 95% exact CI will be provided by dose.

(2) Summary of Overall Response

For overall response, frequency distributions will be provided by dose.

# Statistical/Analytical Issue

### 7.8.4.1 Adjustments for Covariates

Not applicable.

### 7.8.4.2 Handling of Dropouts or Missing Data

Missing test results will not be used for estimations.

For plasma concentrations and laboratory test results, values below the lower limit of quantification will be treated as zero when calculating the descriptive statistics. For laboratory test results, values above the upper limit of quantification will be treated as the upper limit value when calculating the descriptive statistics.

# 7.8.4.3 Multicenter Studies

Not applicable.

### 7.8.4.4 Multiple Comparison/Multiplicity

Not applicable.

### 7.8.4.5 Use of an "Efficacy Subset" of Subjects

Not applicable.

7.8.4.6 Active-Control Studies Intended to Show Equivalence or Non-Inferiority

Not applicable.

7.8.4.7 Examination of Subgroups

Not applicable.

### 7.9

### 7.9.1

### 7.9.1.1 Plasma Concentrations

Analysis Set:

Analysis Variable(s):

Visit:

.arations
.arati

### Analytical Method(s):

The following summaries will be provided by dose.

- (1) Summary of Plasma Concentrations by Visit Descriptive statistics will be provided by visit.
- (2) Mean and Standard Deviation Plot of Plasma Concentrations on Cycle 1 Day 1 and Cycle 1 Day 21

Mean and standard deviation will be plotted. Relative nominal time since last dose (numerical) will be plotted on the horizontal axis and each of the analysis variables will be plotted on the vertical axis for Cycle 1 Day 1 and Cycle 1 Day 21, separately. The vertical axis will be a normal scale.

- (3) Mean Plot of Plasma Concentrations on Cycle 1 Day 1 and Cycle 1 Day 21
  - Mean will be plotted. Relative nominal time since last dose (numerical) will be plotted on the horizontal axis and each of the analysis variables will be plotted on the vertical axis for Cycle 1 Day 1 and Cycle 1 Day 21, separately. The vertical axis will be a common logarithmic scale.
- (4) Plot of Individual Plasma Concentrations on Cycle 1 Day 1 and Cycle 1 Day 21 Individual plasma concentrations will be plotted. Relative actual time since last dose (numerical) will be plotted on the horizontal axis and each of the analysis variables will be plotted on the vertical axis for Cycle 1 Day 1 and Cycle 1 Day 21, separately. The vertical axis will be normal scale.

### 7.9.1.2 Pharmacokinetic Parameters

Analysis Set:

Pharmacokinetic Analysis Set

Analysis Variable(s):

Pharmacokinetic parameters of Niraparib and M1

Cycle 1 Day 1

Cmax, Tmax, AUC24

Cycle 1 Day 21

Cmax, Tmax, AUC24, Cmin, R(AUC24), R(Cmax)

Visit:

Cycle 1 Day 1 and Cycle 1 Day 21

Analytical Method(s):

The following summaries will be provided by dose.

(1) Summary of Pharmacokinetic Parameters by Visit

For Tmax, descriptive statistics will be provided. For other parameters, descriptive statistics, geometric mean, and CV will be provided.

### 7.9.2 Pharmacodynamic Analysis

Not applicable.

### 7.10 Other Outcomes

Not applicable.

### 7.11 Safety Analysis

In this study, safety will be evaluated as the primary endpoint.

### 7.11.1 Adverse Events

7.11.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set:

Safety Analysis Set

Analysis Variable(s):

**TEAE** 

Categories:

Relationship to Study Drug [Related, Not Related]

Analytical Method(s):

The following summaries will be provided by dose.

- (1) Overview of Treatment-Emergent Adverse Events
  - 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects).
  - 2) Relationship of Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects).
  - 3) Grade 3 or higher Treatment-Emergent Adverse Events (number of events, number and percentage of subjects).
  - 4) Grade 3 or higher Drug-Related Treatment-Emergent Adverse Events (number of events, number and percentage of subjects).
  - 5) Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects).
  - 6) Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects).
    - Relationship of serious Treatment-Emergent Adverse Events to study drug (number of events, number and percentage of subjects).
  - 8) Serious Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects).
  - 9) Treatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects).

TEAEs will be counted according to the rules below. Percentages will be based on the number of subjects in the safety analysis set.

### Number of subjects

Summaries for 2) and 7)

and subject to the applicable of Use and Subject to the applicable of Use A subject with occurrences of TEAE in both categories (ie, Related and Not Related) will be counted once in the Related category.

• Summaries other than 2) and 7)

A subject with multiple occurrences of TEAE will be counted only once.

### Number of events

For each summary, the total number of events will be calculated.

7.11.1.2 Frequency of Subjects with DLTs during Cycle 1

Analysis Set:

DLT-evaluable Set

Analysis Variable(s):

DLTs during Cycle 1

Analytical Method(s):

The number and percentage of Subjects with DLTs will be provided by dose.

7.11.1.3 Displays of Treatment-Emergent Adverse events

Analysis Set:

commercial Safety Analysis Set

Analysis Variable(s):

**TEAE** 

Categories:

**Toxicity Grade** 

[Grade 1, Grade 2, Grade 3, Grade 4, Grade 5]

Analytical Method(s):

The following summaries will be provided using frequency distribution by dose.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT.

SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by System Organ Class only or PT only.

- (1) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term.
- (2) Treatment-Emergent Adverse Events by System Organ Class.

- (3) Treatment-Emergent Adverse Events by Preferred Term.
- (4) Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term.
- (5) Toxicity Grade of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term.
- (6) Toxicity Grade of Drug-Related Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term.
- (7) Treatment-Emergent Adverse Events Leading to Study Drug Dose Reduction by System Organ Class and Preferred Term (number of events, number and percentage of subjects).
- (8) Treatment-Emergent Adverse Events Leading to Study Drug Dose Interruption by System Organ Class and Preferred Term (number of events, number and percentage of subjects).
- (9) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term (number of events, number and percentage of subjects).
- (10) Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term.

The frequency distribution will be provided according to the rules below. Percentages will be based on the number of subjects in the safety analysis set.

### Number of subjects

• Summary tables other than (5) and (6)

A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT.

• Summary tables for (5) and (6)

A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum toxicity grade.

# 7.11.1.4 Displays of Pretreatment Events

# Analysis Set:

All Subjects Who Signed the Informed Consent Form

Analysis Variable(s):

**PTE** 

### Analytical Method(s):

PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

(1) Pretreatment Events by System Organ Class and Preferred Term

(2) Serious Pretreatment Events by System Organ Class and Preferred Term

The frequency distribution.

The frequency distribution will be provided according to the rules below.

### Number of subjects

A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only Use only and subject. once in that PT.

## 7.11.2 Clinical Laboratory Evaluations

### 7.11.2.1 Hematology and Serum Chemistry

Analysis Set:

Safety Analysis Set

Analysis Variable(s):

Hematology

Erythrocytes, Hemoglobin, Hematocrit, Platelet Count, Leukocytes with Differentials (ANC, Eosinophils Count, Basophils Count, Absolute Lymphocytes Count, Monocyte Count), MCV

Serum Chemistry

Amylase, Protein (Total Protein), Albumin, ALP, Urea Nitrogen, Creatinine, Magnesium, Total Bilirubin, Sodium, Potassium, Chloride, Calcium, Bicarbonate, Inorganic Phosphate, AST, ALT, LDH, GGT, Glucose (fasted)

Categories:

**Toxicity Grade** [Grade 0, Grade 1, Grade 2, Grade 3, Grade 4]

Cycle 1: Day 1(Predose), Day 8, Day 15

Cycle 2: Day 1, Day 8, Day 15

Cycle 3 and Thereafter: Day 1, Day 8

### Analytical Method(s):

For each variables other than Platelets Count, The following summary (3) will be provided by dose.

For Platelets Count, The following summaries (1)  $\sim$  (3) will be provided by dose.

- (1) Summary of Laboratory Test Results and Change from Baseline by Visit

  Descriptive statistics for observed values and changes from baseline (each postdose visit Predose) will be provided by visit.
- (2) Case Plots of Laboratory Test Results Plots over time for each subject will be presented.
- (3) Summary of Shifts of Laboratory Test Results

Shift tables showing the number of subjects in each category of baseline grade and post-baseline maximum grade for laboratory abnormalities will be provided.

Shift tables showing the number of subjects in each category at Predose and each postdose visit will be provided.

For each laboratory test, the laboratory values will be classified as "Low", "Normal" or "High" relative to the normal reference range. The shift tables will be based on these classifications.

### 7.11.2.2 Urinalysis

Not applicable.

### 7.11.3 Vital Signs and Weight

Not applicable.

### 7.11.4 12-Lead ECGs

Not applicable.

# 7.11.5 Other Observations Related to Safety

Not applicable.

# 7.12 Interim Analysis

Not applicable.

### 7.13 Changes in the Statistical Analysis Plan

From the SAP version 1.0, the following parts were updated. In section 7.1.2, the visit window of clinical laboratory test was modified as below.

Before the change

Section 7.1.2 Definition of Study Visit Windows

Table 7.a Visit Window of Clinical Laboratory Test

| Visit | Scheduled S | | Time Interval (days) Study Day |
|---|---|---|---|
| VISIT | (day | (8) | Study Day |
| Cycle 1, Day 1(Predose) | Study Day: | 1 | - <u>3</u> to 1 |
| Cycle 1, Day 8 | Study Day: | 8 | 5 to 11 |
| Cycle 1, Day 15 | Study Day: | 15 | 12 to 18 |
| Cycle 2, Day 1 | Study Day: | 22 | 19 to 25 |
| Cycle 2, Day 8 | Study Day: | 29 | 26 to 32 |
| Cycle 2, Day 15 | Study Day: | 36 | 33 to 39 |
| Cycle (n) (Cycle 3 and<br>thereafter), Day 1 | Study Day: | 21(n - 1) + 1 | 21(n-1) - 2 to 21(n - 1) + 4 |
| Cycle (n) (Cycle 3 and<br>thereafter), Day 8 | Study Day: | 21(n - 1) + 8 | 21(n - 1) + 5 to 21(n - 1) + 11 |

| | | Scheduled Study Day | | Time Interval (days) |
|---|---|---|---|---|
| Visit | | (days) | | Study Day |
| Cycle 1, Day 1(I | Predose) | Study Day: | 1 | - <u>7</u> to 1 |
| Cycle 1, Da | y 8 | Study Day: | 8 | 5 to 11 |
| Cycle 1, Day | 7 15 | Study Day: | 15 | 12 to 18 |
| Cycle 2, Da | y 1 | Study Day: | 22 | 19 to 25 |
| Cycle 2, Da | y 8 | Study Day: | 29 | 26 to 32 |
| Cycle 2, Day | 7 15 | Study Day: | 36 | 33 to 39 |
| Cycle (n) (Cycle thereafter), D | | Study Day: | 21(n - 1) + 1 | 21(n - 1) - 2 to 21(n - 1) + |
| Cycle (n) (Cycle<br>thereafter), D | | Study Day: | 21(n - 1) + 8 | 21(n - 1) + 5 to 21(n - 1) + |

Properly of Takeda. For non-confine cial use only and subject to the applicable Tames of use